CLINICAL TRIAL: NCT03106519
Title: Distal Extremity (Wrist) Nerve Blocks With a Mixture of Liposome Bupivacaine + Bupivacaine Versus Bupivacaine Alone for Patients Having Dupuytren's Contracture Release: a Blinded Randomized Controlled Trial
Brief Title: Liposome Bupivacaine for WRIST Blocks
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catherine Vandepitte, M.D. (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor-Investigator, Catherine Vandepitte, M.D., Director, New York School of Regional Anesthesia
Organization: New York School of Regional Anesthesia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1601
Record Dates: First submitted 2017-03-24; First posted 2017-04-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Dupuytren's Contracture of the Hand (Viking's Disease)
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single mixture LB & bupivacaine (Experimental): A single mixture of liposome bupivacaine 1.3% (5 mL) + bupivacaine 0.5% (2.5 mL) injected into the median and ulnar nerves
  Interventions: Drug: Liposome bupivacaine + bupivacaine
- Bupivacaine alone (Active Comparator): Bupivacaine 0.5% (7.5 mL) injected into the median and ulnar nerves
  Interventions: Drug: Liposome bupivacaine + bupivacaine

INTERVENTIONS:
Drug: Liposome bupivacaine + bupivacaine

SUMMARY:
Treatment of Dupuytren's contracture requires multiple injections into the palm of the hand to weaken the cords, followed by rupture of the strands 2 days later. Anesthesia is required for both phases of treatment. It is hypothesized that extended-release liposome bupivacaine prolongs nerve blockade of the wrist allowing patients to undergo this 2-part regimen with less pain.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years and max 85 years of age at screening
* Scheduled to undergo Dupuytren's contracture release
* American Society of Anesthesiologists (ASA) physical status I, II or III
* Able to demonstrate sensory function by exhibiting sensitivity to cold, pinprick and light touch
* Female subjects must be surgically sterile or have a monogamous partner who is surgically sterile; at least 2 years postmenopausal; or practicing abstinence; or using an insertable, injectable, transdermal, or combination oral contraceptive approved by the FDA for greater than 2 months prior to screening and commit to the use of an acceptable form of birth control for the duration of the study and for 30 days after completion of the study
* Able to understand the English or Dutch language, purpose and risks of the study
* Able to provide informed consent and authorization to use protected health information, adhere to the study visit schedule and complete all study assessments

Exclusion Criteria:

* Currently pregnant, nursing or planning to become pregnant during the study or within 1 moth after study drug administration
* History of hypersensitivity to local anesthetics
* Contraindication to bupivacaine, paracetamol, ketorolac, oxycodone or morphine
* Medical condition that will make it difficult to assess sensory distributions of peripheral nerves or to communicate with staff
* Chronic scheduled use of any of the following medications within the times specified before surgery: long-acting opioid medication or NSAIDs (except for low-dose aspirin used for cardioprotection) within 3 days, or any opioid medication within 24 hours
* Suspected or known recent history (< 3 months) of drug or alcohol abuse
* Concurrent physical condition that may require analgesic treatment (such as NSAID or opioid) in the postsurgical period for pain that is not strictly related to Dupuytren's contracture and which may confound the postsurgical assessments
* Infection at the planned block site
* Initiation of treatment with any of the following medications within 1 month of study drug administration or if the medication(s) are being given to control pain: selective serotonin reuptake inhibitors (SSRIs), selective norepinephrine reuptake inhibitors (SNRIs), gabapentin, pregabalin (Lyrica®), or duloxetine (Cymbalta®)
* Use of dexmedetomidine HCl (Precedex®) within 3 days of study drug administration
* Body weight <40 kg (88 pounds) or a body mass index >44 kg/m2
* Uncontrolled anxiety, psychiatric, or neurological disorder that might interfere with study assessments
* Any chronic neuromuscular deficit affecting the peripheral nerves or muscles of the surgical extremity
* Any chronic condition or disease that would compromise neurological or vascular assessments
* Presence of preexisting coagulation disorders
* Baseline neurological deficits
* History of impaired kidney function, chronic respiratory disease, rheumatoid arthritis, coagulopathy or loss of sensation in the extremities
* Impaired kidney function (e.g., serum creatinine level >2 mg/dL [176.8 µmol/L] or blood urea nitrogen level >50 mg/dL [17.9 mmol/L]) or impaired liver function (e.g., serum aspartate aminotransferase [AST] level >3 times the upper limit of normal (ULN) or serum alanine aminotransferase [ALT] level >3 times the ULN
* Previous participation in an EXPAREL study
* Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-01-02; Primary Completion 2017-06-28 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Change in current pain over the first postoperative week | From baseline (before nerve block) through first postoperative week
  Pain rating (NRS) at rest and with movement

SECONDARY OUTCOMES:
Change in worst pain over the first postoperative week | From discharge from hospital through first postoperative week
  Modified BRIEF Pain Inventory (Q1)
Change in ability to use hand | From discharge from hospital through first postoperative week
  Hold Styrofoam cup
Change in sleep quality | From discharge from hospital through first postoperative week
  Duration (h), quality rating (0 - 10)
Change in satisfaction with pain control | From discharge from hospital through first postoperative week
  With pain control (0 - 10)
Change in sensory response in skin dermatomes | From beginning of nerve block through first postoperative week
  Cold, pinprick, light touch in the medial and ulnar nerve dermatomes
Change in motor response in thumb and fingers | From beginning of nerve block through first postoperative week
  Abduction/adduction thumb/fingers

OTHER OUTCOMES:
Total number of participants with side effects to regional anesthesia peripheral nerve blockade | From beginning of nerve block through first postoperative week
  Nausea, vomiting, fever, constipation, severe itching of the skin, dizziness, sleepless nights, excessive sweating, urinary retention, headache, heart palpitations
Participants with adverse events | From date of signing ICF through the first postoperative week
  Any untoward medical occurrence (unfavorable and/or unintended change in a body structure or body function) associated with the use of a drug in humans, whether or not considered drug related

CONTACTS AND LOCATIONS:
Overall Officials: Admir Hadzic, MD, PhD, Study Director — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: No